CLINICAL TRIAL: NCT00857103
Title: Improving Patient-Provider Communication in Cancer Care
Brief Title: Effect of Interactive Tailored Assessment on Patient-provider Communication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RCN 177500/V50
Record Dates: First submitted 2009-03-05; First posted 2009-03-06 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-06

CONDITIONS: Lymphoma
Keywords: computer support; patient-provider communication; patient-centered care; cancer
MeSH Terms: conditions — Lymphoma; Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): Standard care
- 2 (Experimental): Use of Choice intervention to support consultations
  Interventions: Behavioral: CHOICE

INTERVENTIONS:
Behavioral: CHOICE — Use of Choice support system as preparation for patient consultations
  Other Names: Standard care
  Arms: 2

SUMMARY:
This interdisciplinary international research collaboration will test effects of Choice, a computer-assisted, interactive support system designed to help cancer patients communicate their symptoms and preferences, and clinicians in incorporating this information into patient care. In this pretest-post test clinical trial with 200 leukemia and lymphoma patients we will: 1) Test effects of Choice when integrated into routine clinical practice on: patient-provider communication, documented patient care, anxiety and patient satisfaction; 2) analyze relationships among the above variables and explore differences in these relationships between groups; 3) analyze group differences in communication style in terms of instrumental and affective behavior, content, participation, initiative and person addressed; and 4) investigate the extent of the time requirements when using Choice in clinical practice, perceived usefulness and ease of use.

DETAILED DESCRIPTION:
Improving shared decision making (SDM), patient-provider communication and incorporating patients' illness experiences and preferences into patient care are high priority health policy goals. However, this is difficult to accomplish without methods and systems that assist patients in sharing their illness experiences and clinicians in integrating this information into patient care. Choice is a computer-assisted, interactive communication and support system for cancer patients designed for this purpose. This interdisciplinary, international research collaboration will test effects of Choice in a pretest-post test clinical trial with 200 leukemia and lymphoma patients. We hypothesize that when patients use Choice for symptom and preference assessments and this information is provided to their clinicians to support consultations in routine practice, (1) patient-provider communication will be more patient-centered; (2) documented care will be more congruent with patients' reported symptoms and preferences; (3) patients will experience lower levels of anxiety and stress during consultations; and (4) they will be more satisfied with the consultation than the "usual care" control group. To better understand the mechanisms by which these effects occur, we will investigate relationships between communication style, documented patient care, anxiety and satisfaction; and explore time requirements, perceived usefulness and ease of use of Choice by patients and clinicians. Controlling for gender, age, diagnosis and type/stage of treatment, analyses of covariance and repeated measurement models will be primarily used for hypotheses testing, correlations and descriptive statistics to answer research questions. This study will contribute to new technologies to support SDM and patient-provider partnerships in health care that can significantly improve patient-provider communication, patient-centered care and physical, emotional and psycho-social well-being of cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with leukemia or lymphoma and in treatment or follow up after treatment within last 12 months.
* Being able to understand, speak and write Norwegian.
* Informed consent

Exclusion Criteria:

* If clinician know patient will receive bad news regarding outcome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2006-08; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | one point assessment
Anxiety | one point assessment
communication | one point assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Rikshospitalet University Hospital, Oslo, Oslo County, Norway

REFERENCES:
- [Derived] Heyn L, Ruland CM, Finset A. Effects of an interactive tailored patient assessment tool on eliciting and responding to cancer patients' cues and concerns in clinical consultations with physicians and nurses. Patient Educ Couns. 2012 Feb;86(2):158-65. doi: 10.1016/j.pec.2011.04.024. Epub 2011 May 17. PMID 21592719